CLINICAL TRIAL: NCT06292650
Title: Prospective, Dose-Escalating, Investigator Initiated Trial to Evaluate the Safety and Efficacy of ZM-02 in Retinitis Pigmentosa
Brief Title: Safety and Efficacy Study of Novel Gene Therapy ZM-02 for Retinitis Pigmentosa Patients
Acronym: MOON
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhongmou Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOON-01
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Retinitis Pigmentosa
Keywords: gene therapy; AAV; RP; optogenetics
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): IVT administration of a single low dose ZM-02 injection
  Interventions: Drug: ZM-02-L
- group 2 (Experimental): IVT administration of a single high dose ZM-02 injection
  Interventions: Drug: ZM-02-H
- group 3 (Sham Comparator): Sham IVT injection
  Interventions: Procedure: ZM-02-S

INTERVENTIONS:
Drug: ZM-02-L — rAAV-PsCatCh2.0 intravitreal injection of low dose
  Other Names: rAAV-PsCatCh2.0e; rAAV-PsCatCh2.0
  Arms: group 1
Drug: ZM-02-H — rAAV-PsCatCh2.0 intravitreal injection of high dose
  Other Names: rAAV-PsCatCh2.0e; rAAV-PsCatCh2.0
  Arms: group 2
Procedure: ZM-02-S — sham intravitreal injection of ZM-02 (not actual injection)
  Other Names: Sham injection
  Arms: group 3

SUMMARY:
This is zM-02's safety, tOlerability, and efficacy in retinitis pigmentOsa first-in-humaN study (MOON). This trial is meant to evaluate the safety and efficacy of ZM-02 in Retinitis pigmentosa (RP) patients. Unilateral intravitreal injections (IVT) will be given into the subject's Study Eye.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is the most common inherited retinal disease. Individuals affected by RP often experience progressive visual impairment, potentially leading to legal blindness. There is currently no established effective clinical treatment available. We developed an innovative adeno-associated virus (AAV)-based gene therapy for individuals with RP, regardless of their causative mutations. Eight to twelve subjects with RP will be recruited and six to nine of them will receive a single unilateral intravitreal injection of ZM-02 at ascending doses, while two to three receive sham injections as the control group.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria can be selected as subjects:

1. Clinically diagnosed with retinal pigment degeneration
2. The visual acuity of study eye is no better than the finger counting, while the visual acuity of the study eye is not better than that of the contralateral eye
3. The subject has had visual experience above the finger counting
4. In the OCT examination of the tested eye, the disappearance of the ellipsoid zone is observed, but the inner nuclear layer and the nerve fiber layer of the retina are still present
5. The refractive power of the tested eye is between -6.00 D and +6.00 D
6. Not infected with the Human Immunodeficiency Virus (HIV) and other acute and chronic infectious diseases
7. Voluntarily sign an Informed Consent Form (ICF), and the age is not less than 18 years and not more than 65 years
8. Able to fully understand and agree to cooperate with the implementation of the research protocol

Exclusion Criteria:

Subjects who meet any one of the following exclusion criteria will be excluded from the study:

1. Pregnant women, breastfeeding women, or male and female subjects who do not agree to contraception during the 12 months before and after medication
2. Subjects with narrow anterior chamber angles or any other medical conditions that contraindicate pupil dilation
3. Subjects allergic to corticosteroids, who are unable to tolerate the corticosteroid treatment described in the protocol, or have active 4. concurrent infections that contraindicate treatment
4. Subjects with systemic diseases, or other medical or mental illnesses, or other safety concerns for the study
5. Subjects with other symptoms and/or diseases or conditions that can alter visual function, including but not limited to glaucoma and central nervous system lesions (mild cataracts are not included in this restriction)
6. Eye diseases that may interfere with the assessment of vision during the study and/or interfere with other ocular assessments such as OCT
7. Diseases that may affect the clinical trial, such as tumors, metabolic, immune-related diseases, etc.
8. Subjects who have undergone major eye surgery within the last 3 months before screening
9. Subjects with a history of malignant tumors within the last 5 years
10. Subjects with other retinal diseases not suitable for this study, such as retinal detachment
11. Patients undergoing or potentially undergoing immunosuppressive treatment for other diseases, excluding this study
12. Participation in any clinical trials other than this study within the last 3 months
13. Subjects who have received gene therapy outside of this study
14. Other reasons deemed by the researcher as unsuitable for participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2027-12-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | baseline to day 3, week 1, 4, 12, 24, 36, 52
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that leading to the following: Results in death; Life-threatening, refers to an event in which the patient is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe; Significant or permanent disability/incapacity, where disability refers to a serious disruption and damage of a person's ability to perform normal life functions; Requires inpatient hospitalization or prolongation of existing hospitalization; Congenital anomaly or birth defect; Other medically important events.
Changes in intraocular pressure (IOP) in Subjects | baseline to day 3, week 1, 4, 12, 24, 36, 52
  IOP refers to the fluid pressure inside the eye. Monitoring IOP ensures that interventions do not inadvertently increase IOP to dangerous levels. IOP will be measured using a clinical tonometry device.

SECONDARY OUTCOMES:
Change of MLMT level | baseline to day 3, week 1, 4, 12, 24, 36, 52
  Multi-Luminance Mobility Test (MLMT) is used to evaluate how well individuals with visual impairments can navigate and perform tasks in different lighting conditions. This test is particularly relevant for conditions that affect night vision or light adaptation, such as retinitis pigmentosa or other forms of inherited retinal dystrophies.
Change of Quality of Life | baseline to day 3, week 1, 4, 12, 24, 36, 52
  Quality of Life will be measured using Visual Function Questionnaire (VFQ-25) or other similar questionnaires before and after treatment
Change in best corrected visual acuity (BCVA) | baseline to day 3, week 1, 4, 12, 24, 36, 52
  BCVA of both eyes will be assessed using the early treatment of diabetic retinopathy study (ETDRS) chart or tumbling "E" chart or other avaliable measurement. This approach was chosen to facilitate visual acuity testing in subject who cannot recognize letters.

OTHER OUTCOMES:
Change in color discrimination | baseline to day 3, week 1, 4, 12, 24, 36, 52
  Color discrimination testing measures an individual's ability to perceive and differentiate hues across the visible spectrum under standard luminance level. Instead of relying on fine spatial detail, these tests challenge the visual system to detect subtle differences in wavelength-an ability that is often impaired in advanced retinal disease.
Change in visual field (VF) | baseline to day 3, week 1, 4, 12, 24, 36, 52
  Visual field will be assessed by Humphrey perimetry, changes in VFI, MD, PSD will be analyzed.
Change in Fundus Autofluorescence (FAF) | baseline to day 3, week 1, 4, 12, 24, 36, 52
  FAF is a non-invasive imaging technique that provides critical information about the health of the retina, which is vital for the functioning of the retina.
Change in central foveal thickness (CFT) using Optical Coherence Tomography (OCT) | baseline to day 3, week 1, 4, 12, 24, 36, 52
  Central Foveal Thickness refers to the thickness of the retina at the fovea, the central part of the macula. Changes in CFT can indicate various retinal conditions, including macular edema, macular degeneration, and central serous retinopathy.
Change in central macular thickness (CMT) using Optical Coherence Tomography (OCT) | baseline to day 3, week 1, 4, 12, 24, 36, 52
  Central Macular Thickness is the measurement of the thickness of the macula, which includes the fovea and the small surrounding area. The macula is responsible for central vision and visual acuity.
Changes in the fundus using fundus color photography | baseline to day 3, week 1, 4, 12, 24, 36, 52
  Fundus photography is used to document and monitor changes in the eye over time. It's vital for assessing the conditions of retina and monitoring the effects of treatments.
Change of MLCBT level | baseline to day 3, week 1, 4, 12, 24, 36, 52
  Multi-luminance chess board test (MLCBT) is a functional vision assessment specifically designed for individuals with severe visual impairment. During the test, participants are asked to identify the orientation of light target and avoid chessboard pattern obstacles presented under multiple illumination levels that simulate real-world environments, from very dim to bright light conditions. By evaluating performance across luminance tiers, MLCBT provides a sensitive measure of residual spatial vision and contrast-dependent functional gains, enabling the detection of clinically meaningful improvements that are not captured by conventional visual acuity testing.
Change of MLSDT level | baseline to day 3, week 1, 4, 12, 24, 36, 52
  The Multi-Luminance Shape Discrimination Test (MLSDT) evaluates functional vision by measuring a participant's ability to recognize geometric shapes presented at high contrast under different luminance levels. Shapes such as circles, squares, or triangles are shown one at a time, and the participant must correctly identify each target. By testing performance across a range of light intensities that mimic everyday environments, MLSDT sensitively captures changes in spatial perception and object recognition. This makes it particularly valuable for assessing treatment-related improvements in individuals with profound vision loss, where traditional acuity metrics may not reflect meaningful functional gains.
Change of FST outcome | baseline to day 3, week 1, 4, 12, 24, 36, 52
  The Full Stimulus Test (FST) is a test to assess the functional integrity of the entire visual pathway, from the retina to the visual cortex. It often used in studies involving retinal dystrophies or certain neuro-ophthalmological conditions, FST might be used to assess the efficacy of a treatment or intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wei, PhD, Principal Investigator — Beijing Tongren Hospital, CMU
Locations (1):
- Beijing Tongren Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No